CLINICAL TRIAL: NCT01489059
Title: A Phase I Dose Escalation Study of BMS-982470 (Recombinant Interleukin 21, rIL-21) in Combination With Ipilimumab in Subjects With Unresectable Stage III or Stage IV Melanoma
Brief Title: Safety Study of IL-21/Ipilimumab Combination in the Treatment of Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA220-007
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1 - Arm 1: BMS-982470 (Daily x 5) + Ipilimumab (Experimental): Dose Escalation
  Interventions: Biological: BMS-982470 (recombinant interleukin-21); Biological: Ipilimumab
- Part 1 - Arm 2: BMS-982470 (Weekly) + Ipilimumab (Experimental): Dose Escalation
  Interventions: Biological: BMS-982470 (recombinant interleukin-21); Biological: Ipilimumab
- Part 2 - Arm 1: BMS-982470 (Daily x 5) + Ipilimumab (Experimental): Cohort Expansion
  Interventions: Biological: BMS-982470 (recombinant interleukin-21); Biological: Ipilimumab
- Part 2 - Arm 2: BMS-982470 (Weekly) + Ipilimumab (Experimental): Cohort Expansion
  Interventions: Biological: BMS-982470 (recombinant interleukin-21); Biological: Ipilimumab
- Part 2 - Arm 3: Ipilimumab monotherapy (Active Comparator): Cohort Expansion
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: BMS-982470 (recombinant interleukin-21) — Solution, Intravenous, 10,30,50 μg/kg, daily for 5 days every 3 weeks (daily x 5), 16-20 weeks depending on response
  Arms: Part 1 - Arm 1: BMS-982470 (Daily x 5) + Ipilimumab
Biological: BMS-982470 (recombinant interleukin-21) — Solution, Intravenous, 30,100,150 μg/kg, weekly, 16-20 weeks depending on response
  Arms: Part 1 - Arm 2: BMS-982470 (Weekly) + Ipilimumab
Biological: BMS-982470 (recombinant interleukin-21) — Solution, Intravenous, Maximum tolerated dose from Part 1, daily for 5 days every 3 weeks (daily x 5), 12-16 weeks depending on response
  Arms: Part 2 - Arm 1: BMS-982470 (Daily x 5) + Ipilimumab
Biological: BMS-982470 (recombinant interleukin-21) — Solution, Intravenous, Maximum tolerated dose from Part 1, Weekly, 12-16 weeks depending on response
  Arms: Part 2 - Arm 2: BMS-982470 (Weekly) + Ipilimumab
Biological: Ipilimumab — Solution, Intravenous, 1,3,10 mg/kg, every 3 weeks, 16-20 weeks depending on response
  Other Names: Yervoy®
  Arms: Part 1 - Arm 1: BMS-982470 (Daily x 5) + Ipilimumab; Part 1 - Arm 2: BMS-982470 (Weekly) + Ipilimumab
Biological: Ipilimumab — Solution, Intravenous, Maximum tolerated dose from Part 1, every 3 weeks, 12-16 weeks depending on response
  Other Names: Yervoy®
  Arms: Part 2 - Arm 1: BMS-982470 (Daily x 5) + Ipilimumab; Part 2 - Arm 2: BMS-982470 (Weekly) + Ipilimumab
Biological: Ipilimumab — Solution, Intravenous, 3mg/kg, Every 3 weeks, 12-16 weeks depending on response
  Other Names: Yervoy®
  Arms: Part 2 - Arm 3: Ipilimumab monotherapy

SUMMARY:
The purpose of this study is to determine whether the combination of interleukin-21 (IL-21) and Ipilimumab in subjects with melanoma is safe, and provide preliminary information on the clinical benefits of the combination compared with Ipilimumab alone

DETAILED DESCRIPTION:
Allocation: Part 1 Dose Escalation Phase: Non-randomized; Part 2 Cohort Expansion Phase: Randomized

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Unresectable Stage III or Stage IV melanoma
* Part 1 Dose Escalation: Prior melanoma treatment allowed except for the following: ipilimumab, BMS-982470 (rIL-21), anti-Programmed Death-1 (anti-PD-1), anti-programmed death-ligand 1 (anti-PD-L1), anti-PD-L2 or anti-CD137
* Part 2 Cohort expansion: Prior treatment for melanoma is not allowed, except for adjuvant therapy with interferon alpha or melanoma vaccines which are permitted
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI)
* Normal liver function tests

Exclusion Criteria:

* Part 1 Dose escalation: subjects with ≤ 2 brain metastases of stable size, ≥ 4 weeks post-radiation treatment, and off steroids are allowed
* Part 2 Cohort expansion: subjects with known or suspected brain metastases and uveal melanoma are excluded
* Autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Part1 (Dose Escalation): The Maximum tolerated dose (MTD) of BMS-982470 using 2 distinct schedules when administered in combination with Ipilimumab | Within the first 63 days
  Based on the dose-limiting toxicity (DLT) rate
Part 2 (Cohort Escalation): Safety and tolerability of the MTD dose for each of the schedules | 84 days on treatment
  Based on medical review of AE reports and the results of vital sign measurements, physical examinations, medical history, and clinical laboratory tests

SECONDARY OUTCOMES:
Efficacy of BMS-982470 in combination with Ipilimumab as measured by objective response | Baseline (Day 1), End of Treatment (EOT) [3 weeks after last dose of Ipilimumab], 3 and 6 months Follow-up
Area under the serum concentration-time curve from time zero to the last quantifiable concentration [AUC(0-T)] of BMS-982470 and Ipilimumab | 20 time points during Lead-In Cycle; Up to 11 time points during Cycle 3
Area under the serum concentration-time curve in one dosing interval [AUC(TAU)] of BMS-982470 and Ipilimumab | 20 time points during Lead-In Cycle; Up to 11 time points during Cycle 3
Area under the serum concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] of BMS-982470 and Ipilimumab | 20 time points during Lead-In Cycle; Up to 11 time points during Cycle 3
The maximum observed serum concentration (Cmax) of BMS-982470 and Ipilimumab | 20 time points during Lead-In Cycle; Up to 11 time points during Cycle 3
Trough observed serum concentration (Cmin) of BMS-982470 and Ipilimumab | 1 time point each 3-week Cycle
The time of maximum observed serum concentration (Tmax) of BMS-982470 and Ipilimumab | 20 time points during Lead-In Cycle; Up to 11 time points during Cycle 3
Serum half-life (T-HALF) of BMS-982470 and Ipilimumab | 20 time points during Lead-In Cycle; Up to 11 time points during Cycle 3
Apparent total body clearance (CLT) of BMS-982470 and Ipilimumab | 20 time points during Lead-In Cycle; Up to 11 time points during Cycle 3
Apparent volume of distribution at steady state (Vss) of BMS-982470 and Ipilimumab | 20 time points during Lead-In Cycle; Up to 11 time points during Cycle 3
Incidence of BMS-984270 and Ipilimumab Anti-Drug Antibodies | Up to 6 months following last dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (9):
- United States (8):
  - Oncology Research Associates, Pllc D/B/A, Scottsdale, Arizona
  - Ucla Hematology/Oncology., Los Angeles, California
  - H. Lee Moffitt Cancer Center & Research Inst, Inc, Tampa, Florida
  - Indiana University Health Melvin And Bren Simon Cancer Center, Indianapolis, Indiana
  - University Of Louisville Medical Center, Inc., Dba, Louisville, Kentucky
  - Portland Providence Medical Center, Portland, Oregon
  - Md Anderson Can Cnt, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Local Institution, San Juan, Puerto Rico

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx